CLINICAL TRIAL: NCT06464692
Title: A Phase 1b Study to Evaluate Safety and Pharmacokinetics (PK) of Telisotuzumab Adizutecan (ABBV-400) in Chinese Subjects With Unresectable Locally Advanced/Metastatic Colorectal Cancer
Brief Title: Study to Assess Adverse Events and How Intravenously (IV) Infused Telisotuzumab Adizutecan (ABBV-400) Moves Through the Body of Adult Participants With Unresectable Locally Advanced/Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M24-559
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; CRC; Telisotuzumab Adizutecan (ABBV-400); Unresectable Locally Advanced/Metastatic CRC
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Safety Run-In Cohort 1: Telisotuzumab Adizutecan Dose A (Experimental): Participants with unresectable locally advanced/metastatic colorectal cancer (CRC) will receive telisotuzumab adizutecan dose A during the approximately 2.5 year study duration.
  Interventions: Drug: Telisotuzumab Adizutecan
- Safety Run-In Cohort 2: Telisotuzumab Adizutecan Dose B (Experimental): Participants with unresectable locally advanced/metastatic CRC will receive telisotuzumab adizutecan dose B during the approximately 2.5 year study duration.
  Interventions: Drug: Telisotuzumab Adizutecan
- Dose Expansion Part 1: Telisotuzumab Adizutecan Dose A (Experimental): Participants with unresectable locally advanced/metastatic CRC will receive telisotuzumab adizutecan dose A during the approximately 2.5 year study duration.
  Interventions: Drug: Telisotuzumab Adizutecan
- Dose Expansion Part 2: Telisotuzumab Adizutecan Dose C (Experimental): If further analysis is warranted, participants with unresectable locally advanced/metastatic CRC will receive telisotuzumab adizutecan dose C during the approximately 2.5 year study duration.
  Interventions: Drug: Telisotuzumab Adizutecan

INTERVENTIONS:
Drug: Telisotuzumab Adizutecan — Intravenous (IV) Infusion

SUMMARY:
Colorectal cancer (CRC) is the third most common type of cancer diagnosed worldwide and in China. The purpose of this study is to assess adverse events and how telisotuzumab adizutecan moves through the body of adult participants with unresectable locally advanced/metastatic CRC.

Telisotuzumab adizutecan is an investigational drug being developed for the treatment of CRC. Study doctors put the participants in cohorts called treatment arms. Each treatment arm receives a different dose of telisotuzumab adizutecan. This study will include a dose escalation phase followed by a dose expansion phase. Up to approximately 30 adult participants with unresectable locally advanced/metastatic CRC, will be enrolled in the study in approximately 8 sites in China.

In the dose escalation arms, participants will receive escalating doses of intravenously (IV) infused telisotuzumab adizutecan dose A or B. In dose expansion arm part 1, participants will receive dose A of IV infused telisotuzumab adizutecan. In dose expansion arm part 2, participants will receive the dose C of IV infused telisotuzumab adizutecan. The total study duration will be approximately 2.5 years.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests, questionnaires and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1.
* Has histologically or cytologically confirmed unresectable advanced/metastatic colorectal cancer (mCRC).
* Has measurable disease per response evaluation criteria in solid tumors (RECIST) v1.1.
* Does not harbor the BRAF V600E mutation and is not deficient mismatch repair (dMMR)+/microsatellite instability (MSI)-High.
* Stage 2 only:

  * Archival or recently obtained tumor material must be submitted for assessment of c-Met protein levels by an AbbVie designated IHC laboratory during the pre-screening period. Tumor material from the primary tumor site and/or metastatic sites are allowed. If archival tissue is negative for c-Met protein expression with 3+ intensity, >= 10% tumor cells, recently obtained biopsy material may be submitted for reassessment of c-Met protein expression with 3+ intensity, >= 10% tumor cells.

Exclusion Criteria:

* History (within 6 months) of congestive heart failure (defined as New York Heart Association, Class 2 or higher), ischemic cardiovascular event, cardiac arrhythmia requiring pharmacological or surgical intervention, pericardial effusion, or pericarditis.
* Prior systemic regimen containing c-Met protein targeting antibody (e.g., amivantamab-vmjw, ABT-700) or define: antibody-drug conjugate (ADC). Tyrosine kinase inhibitors (TKIs) of Met protein are allowed.
* History of Interstitial lung disease (ILD)/pneumonitis that required treatment with systemic steroids, or any evidence of active ILD/pneumonitis on screening chest computed tomography (CT) scan.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis.
* History of clinically significant, intercurrent lung-specific illnesses including, but not limited to:

  * Underlying pulmonary disorder (i.e., pulmonary emboli within 3 months of the study enrollment, severe asthma, severe chronic obstructive pulmonary disease [COPD], restrictive lung disease, pleural effusion, dependence on supplemental oxygen, etc.)
  * Any autoimmune, connective tissue or inflammatory disorders with documented or suspicious pulmonary involvement at screening (i.e., rheumatoid arthritis, Sjogren's, sarcoidosis, etc.) and prior pneumonectomy.
* No resolution of any acute clinically significant treatment-related toxicity from prior therapy to Grade <= 1 prior to study entry, except for neutropenia (Grade <= 2), peripheral neuropathy (Grade <= 2), and alopecia (any grade).
* Untreated brain or meningeal metastases (i.e., participants with history of metastases are eligible provided they do not require ongoing steroid treatment for cerebral edema and have shown clinical and radiographic stability for at least 14 days after definitive therapy).
* History of other malignancies within 5 years prior to screening, except for malignancies with a negligible risk of metastasis or death (e.g., 5-year Overall Survival [OS] rate > 90%).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) of Telisotuzumab Adizutecan in Stage 1 | Up to 24 Months
  DLTs are defined as grade >= 3 thrombocytopenia that cannot clinically improve after adequate medical treatment/support, febrile neutropenia grade >= 3 or grade 4 neutropenia that cannot clinically improve after adequate medical treatment/support, and any grade 2 or higher interstitial lung disease (ILD)/pneumonitis that cannot clinically improve after adequate medical treatment/support.
Maximum observed plasma or serum concentration (Cmax) of Telisotuzumab Adizutecan Conjugate | Up to 24 Months
  Cmax of telisotuzumab adizutecan conjugate.
Time to Cmax (Tmax) of Telisotuzumab Adizutecan Conjugate | Up to 24 Months
  Tmax of telisotuzumab adizutecan conjugate.
Area Under the Concentration-Time Curve (AUC) of Telisotuzumab Adizutecan Conjugate | Up to 24 Months
  AUC of telisotuzumab adizutecan conjugate.
Total Antibody of Telisotuzumab Adizutecan | Up to 24 Months
  Total antibody of telisotuzumab adizutecan.
Unconjugated Payload of Telisotuzumab Adizutecan | Up to 24 Months
  Unconjugated payload of telisotuzumab adizutecan.

SECONDARY OUTCOMES:
Objective Response (OR) | Up to 24 Months
  OR as assessed by the Investigator: Confirmed complete response (CR) or confirmed partial response (PR) as assessed by the Investigator per Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1.
Duration of Response (DoR) | Up to 24 Months
  DoR as assessed by Investigator: DoR is defined as the time from the participantt's initial response (CR or PR) to the first occurrence of radiographic progression or death from any cause.
Best Overall Response (BOR) | Up to 24 Months
  Disease control as assessed by the Investigator: BOR of confirmed CR or confirmed PR, or stable disease based on RECIST, version 1.1.
Progression-Free Survival (PFS) | Up to 24 Months
  PFS as assessed by Investigator: PFS is defined as the time from the participant's first dose of study treatment until radiographic progression or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to 24 Months
  OS is defined as the time from the participant's first dose of study treatment until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (8):
- China (8):
  - Beijing Cancer Hospital /ID# 263297, Beijing, Beijing Municipality
  - The Sixth Affiliated Hospital of Sun Yat-sen University /ID# 263309, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital /ID# 263049, Harbin, Heilongjiang
  - Henan Cancer Hospital /ID# 263172, Zhengzhou, Henan
  - Hubei Cancer Hospital /ID# 263248, Wuhan, Hubei
  - The First Affiliated Hospital of Nanchang University /ID# 263193, Nanchang, Jiangxi
  - First Affiliated Hospital of China Medical University /ID# 263338, Shenyang, Liaoning
  - The Second Affiliated Hospital of Zhejiang University School of Medicine /ID# 263094, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-559